CLINICAL TRIAL: NCT03111940
Title: The Oxford Optimisation of PCI Study (OXOPT-PCI Study)
Acronym: OXOPT-PCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Adrian Banning, Professor, Oxford University Hospitals NHS Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12005
Record Dates: First submitted 2016-06-12; First posted 2017-04-13 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

ARMS (2):
- PCI optimisation (Experimental): Post PCI FFR below 0.9
  Interventions: Procedure: Optimisation of the result of intracoronary stenting according to specific algorithm
- No PCI optimisation (No Intervention): Post PCI FFR 0.9 or higher

INTERVENTIONS:
Procedure: Optimisation of the result of intracoronary stenting according to specific algorithm
  Arms: PCI optimisation

SUMMARY:
The OxOPT-PCI study addresses patients with coronary artery disease who are referred to the John Radcliffe Hospital because of the need for treatment with an intra-coronary stent (metal scaffold) for clinical reasons. Although, this has become a highly standardised procedure it is still challenging for the clinician to assess the final success of this procedure at the end of intervention with conventional methods. This shortcoming can potentially translate into a worse clinical outcome for approximately 10 percent of all patients treated with an intra-coronary stent for this type of disease.

This study (OxOPT-PCI) investigates if the use of blood flow measurements (namely measurement of fractional flow reserve (FFR)) and intravascular imaging (namely optical coherence tomography (OCT)) after the implantation of a stent can improve the treatment result for these patients. Both, FFR and OCT are being used already in daily clinical routing but their usefulness especially in combination is not clear. In order to standardise the optimisation procedure we developed a specific algorithm to make sure that all patients receive the same optimisation measures based on the assessment of FFR and OCT.

The benefit of this specific optimisation algorithm will be assessed by measuring 1) indices of coronary blood flow, 2) intravascular imaging at the end of the procedure, and 3) by contacting the patients 12 months after stenting to verify the clinical mid-term success.

ELIGIBILITY:
Inclusion Criteria:

* participant is willing and able to give informed consent for participation in the study
* angiogram shows haemodynamically relevant lesion suitable for PCI and suitable for the use of intravascular imaging (OCT)

Exclusion Criteria:

* patients in whom safety or clinical concerns preclude participation
* ST-segment elevation myocardial infarction
* presentation with cardiogenic shock
* revascularization by mean of balloon angioplasty without stenting
* contraindications to adenosine

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospital - NHS Trust, Oxford, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible subjects were referred for elective or urgent complex PCI between September 2016 and July 2017 at the John Radcliffe Hospital, Oxford Heart Centre, United Kingdom. All patients underwent conventional angiography-guided stent deployment, until an acceptable angiographic result was achieved. Following completion of conventional PCI, FFR was measured, and intracoronary OCT imaging was performed. The study population was then divided into two groups based on the observed FFR value.
Pre-assignment Details: 35 pts recruited
Groups:
- Group 1 Patients With a Suboptimal Functional Result (FFR <0.90) After Conventional PCI: OCT was performed per protocol after achievement of satisfactory angiographic results. OCT was analysed according to the presence of one or more of the following according to CLI-OPCI study criteria: stent underexpansion and/or incomplete lesion coverage and/or stent malapposition and/or stent-edge dissection and/or intra-stent plaque/thrombus protrusion. Operators were mandated to perform PCI optimisation according to the respective OCT finding.
- Group 2 Patients With a Satisfactory Functional Result (FFR ≥0.90) After Conventional PCI: No further PCI optimisation was performed and OCT acquisition was performed only as a safety measure, to assess the frequency of relevant vessel-related complications
Period: Overall Study
Arm/Group | Group 1 Patients With a Suboptimal Functional Result (FFR <0.90) After Conventional PCI | Group 2 Patients With a Satisfactory Functional Result (FFR ≥0.90) After Conventional PCI
Started | 21 | 14
Completed | 21 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1 Patients With a Suboptimal Functional Result (FFR <0.90) After Conventional PCI: In patients in Group 1, OCT was performed per protocol after achievement of satisfactory angiographic results. OCT was analysed according to the CLI-OPCI study defining a suboptimal stent result according to specific criteria. For patients that fulfilled OCT criteria for optimisation (Group 1A), operators were mandated to perform PCI optimisation according to the respective OCT finding. For patients in Group 1 who did not fulfil the OCT criteria (Group 1B), further PCI optimisation was not performed.
- Group 2 Patients With a Satisfactory Functional Result (FFR ≥0.90) After Conventional PCI: For patients in Group 2, no further PCI optimisation was performed and OCT acquisition was performed only as a safety measure, to assess the frequency of relevant vessel-related complications.
- Total: Total of all reporting groups
Arm/Group | Group 1 Patients With a Suboptimal Functional Result (FFR <0.90) After Conventional PCI | Group 2 Patients With a Satisfactory Functional Result (FFR ≥0.90) After Conventional PCI | Total
Number analyzed (Participants) | 21 | 14 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (8.4) | 64.8 (8.2) | 64.4 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 18 | 11 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 14 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 21 | 14 | 35

OUTCOME MEASURES:

1. Primary Outcome: Final Fractional Flow Reserve (FFR) After Intracoronary Stenting
Description: After administration of intracoronary nitrates, FFR was measured under maximal hyperaemia, using intravenous adenosine (140 mg kg-1 min-1) as the ratio between distal coronary pressure (Pd) and aortic pressure (Pa)
Time Frame: Immediately post-stenting for Group 1A and 1B, and post FFR/OCT-guided optimisation for Group 1A
Population: OCT-guided PCI optimisation was only performed in Group 1A
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Group 1A: OCT-guided PCI Optimisation: Patients from Group 1 who fulfilled the OCT criteria and further PCI optimisation was performed
- Group 1B: No PCI Optimisation Performed: Patients from Group 1 who did not fulfil the OCT criteria, and thus, further PCI optimisation was not performed
Arm/Group | Group 1A: OCT-guided PCI Optimisation | Group 1B: No PCI Optimisation Performed
Number analyzed (Participants) | 13 | 8
Ratio
  Immediately post-stenting | 0.80 (0.02) | 0.84 (0.03)
  Post OCT-guided optimisation: number analyzed (Participants) | 13 | 0
  Post OCT-guided optimisation | 0.88 (0.01) |

2. Secondary Outcome: Number of Participants With Stent-edge Dissection Assessed by OCT
Description: Defined as presence of a linear rim of tissue ≥200 μm in width and with clear separation from the vessel wall, or underlying plaque <5 mm from stent edges
Time Frame: During PCI procedure, OCT typically adds 5 minutes to the procedure
Measure: Count of Participants; unit: Participants
Groups:
- Group 1A: Post-stenting FFR Below 0.9, FFR/OCT Optimisation Performed: OCT fulfilled optimisation criteria Presence of one or more of the following criteria for optimisation: stent underexpansion and/or incomplete lesion coverage and/or stent malapposition and/or stent-edge dissection and/or intra-stent plaque/thrombus protrusion.
- Group 2: Post-stenting FFR 0.9 or Higher: No further PCI optimisation performed and OCT acquisition performed only as safety measure to assess frequency of relevant vessel-related complications
Arm/Group | Group 1A: Post-stenting FFR Below 0.9, FFR/OCT Optimisation Performed | Group 2: Post-stenting FFR 0.9 or Higher
Number analyzed (Participants) | 13 | 14
Participants | 2 | 1

3. Secondary Outcome: Number of Participants With Reference Lumen Narrowing (Geographical Miss) Assessed by OCT
Description: Defined as reference lumen area <4.5 mm2, with significant residual plaque within 10 mm of stent edges
Time Frame: During PCI procedure, OCT typically adds 5 minutes to the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1A: Post-stenting FFR Below 0.9, FFR/OCT Optimisation Performed | Group 2: Post-stenting FFR 0.9 or Higher
Number analyzed (Participants) | 13 | 14
Participants | 5 | 0

4. Secondary Outcome: Number of Participants With Stent Malapposition Assessed by OCT
Description: Defined as stent-adjacent vessel lumen distance > 200 μm
Time Frame: During PCI procedure, OCT typically adds 5 minutes to the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1A: Post-stenting FFR Below 0.9, FFR/OCT Optimisation Performed | Group 2: Post-stenting FFR 0.9 or Higher
Number analyzed (Participants) | 13 | 14
Participants | 7 | 3

5. Secondary Outcome: Number of Participants With Plaque/Thrombus Protrusion Assessed by OCT
Description: Defined as tissue prolapsing between stent struts extending inside a circular arc connecting adjacent struts or intraluminal mass ≥500 μm thick with no direct connection to the vessel wall, or highly backscattered luminal protrusion in continuity with the vessel wall, resulting in signal-free shadowing
Time Frame: During PCI procedure, OCT typically adds 5 minutes to the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1A: Post-stenting FFR Below 0.9, FFR/OCT Optimisation Performed | Group 2: Post-stenting FFR 0.9 or Higher
Number analyzed (Participants) | 13 | 14
Participants | 1 | 1

6. Secondary Outcome: Number of Participants With Stent Under-expansion Assessed by OCT
Description: Defined as minimal stent area (MSA) < 70% of average reference lumen area and/or MSA < 4.5 mm2
Time Frame: During PCI procedure, OCT typically adds 5 minutes to the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1A: Post-stenting FFR Below 0.9, FFR/OCT Optimisation Performed | Group 2: Post-stenting FFR 0.9 or Higher
Number analyzed (Participants) | 13 | 14
Participants | 6 | 0

ADVERSE EVENTS:
Time Frame: During procedure, approximately 1 hour and 30 minutes
Groups:
- PCI Optimisation: Post PCI FFR below 0.9
  Optimisation of the result of intracoronary stenting according to specific algorithm
Arm/Group | PCI Optimisation | No PCI Optimisation
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/14
Other Adverse Events (participants affected / at risk) | 0/21 | 0/14

LIMITATIONS AND CAVEATS:
Small sample size and non-randomized observational nature limiting statistical power; Larger randomised trials are required to determine clinical impact of any final combined imaging/physiology assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2016-09-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT03111940/Prot_000.pdf